CLINICAL TRIAL: NCT02971267
Title: Follow-up of the Inflammatory Cardiomyopathy Cohort of SFB/TR19
Brief Title: Follow-up of the Cardiomyopathy Cohort SFB/TR19
Acronym: SFB/TR19plus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: SFB/TR19plus-001
Record Dates: First submitted 2016-11-09; First posted 2016-11-22 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Cardiomyopathies; Heart Failure
Keywords: heart failure; cardiomyopathy; myocarditis
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Myocarditis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational — None, observational only

SUMMARY:
Follow-up of a cohort of inflammatory cardiomyopathy patients (suspected or validated inflammatory cardiomyopathy) recruited at baseline by the SFB-TR19 project. Standardized protocols will be used for the assessment of medical history and examinations, laboratory biomarkers, and the collection of various biomaterials for biobanking purposes.

DETAILED DESCRIPTION:
Periodical follow-up of a cohort of inflammatory cardiomyopathy patients (suspected or validated inflammatory cardiomyopathy) recruited at baseline by the SFB/TR19 project. Participants will be followed up at least every year - or more frequently based on clinical need. Standardized protocols will be used for the assessment of medical history and examinations, laboratory biomarkers, and the collection of various biomaterials for biobanking purposes.

ELIGIBILITY:
Inclusion Criteria:

* Participation in baseline examination of SFB/TR19

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or validated inflammatory cardiomyopathy at baseline
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-06; Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular events | 1-year follow-ups up to 10 years
  Number of hospitalization (HF based. all-cause), interventions (ICD, pacemaker), myocardial infarction

SECONDARY OUTCOMES:
LVEF (left ventricular ejection fraction) | 1-year follow-ups up to 10 years
  Left ventricular ejection fraction at time of follow-ups (through study completion, every year)
VO2peak | 1-year follow-ups up to 10 years
  Exercise capacity by CPET (cardiopulmonary exercise testing)
QOL | 1-year follow-ups up to 10 years
  Quality of life by MLHF questionnaire
Mortality | 1-year follow-ups up to 10 years
  Mortality (HF-related, cardiovascular disease, all-cause mortality)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine B, University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No